CLINICAL TRIAL: NCT05750550
Title: Acute Effect of Instrument-Assisted Soft Tissue Mobilization on Hamstring Flexibility Via Fascial Chain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GaziosmanpasaU_Erol_06
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Instrument Assisted Soft Tissue Mobilization Group (Experimental): With the IASTM device, application will be made over the skin to the triceps surae muscle and plantar fascia for 15 minutes. The application will be made in the prone position. Massage oil will be used to reduce tissue friction before the application.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — With the IASTM device, application will be made over the skin to the triceps surae muscle and plantar fascia for 15 minutes. The application will be made in the prone position. Massage oil will be used to reduce tissue friction before the application.

SUMMARY:
Instrument assisted soft tissue mobilization (IASTM) is one of the methods used to achieve fascial release. In this study, it will be examined whether there will be an increase in hamstring flexibility by releasing the superficial posterior fascial chain as a result of the IASTM technique to be applied over the triceps surae muscle and plantar fascia. Sociodemographic information of individuals who meet the inclusion criteria and volunteer to participate in the study will be obtained, and straight leg lift test and popliteal angle measurement will be performed with the digital inclinometer (Baseline Digital Inclinometer) to be provided within the scope of the project to measure hamstring flexibility. Then, IASTM will be applied to the triceps surae muscle and plantar fascia for 15 minutes. Measurements will be repeated after the application.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with a straight leg lift test less than 80° and a popliteal angle greater than 15° will be included in the study.

Exclusion Criteria:

* Individuals with a history of lower extremity fractures, lumbar disc herniation, acute pain, a history of lesion in the hamstring muscles at least 1 month before the study, knee or hip prosthesis, and those using drugs that may affect the measurements (e.g., muscle relaxants) will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Straight Leg Raise Test | Baseline
  Measurements will be made with a digital inclinometer. In the supine position, the digital inclinometer will be inserted into the tuberositas tibia. Then, the participant's leg will be passively lifted by the researcher with the knee extended. The leg will be brought to the point where the tension is felt, where the value on the inclinometer will be recorded. It will then return to the starting position. The procedure will be repeated for both legs.
Straight Leg Raise Test | 1 hour
  Measurements will be made with a digital inclinometer. In the supine position, the digital inclinometer will be inserted into the tuberositas tibia. Then, the participant's leg will be passively lifted by the researcher with the knee extended. The leg will be brought to the point where the tension is felt, where the value on the inclinometer will be recorded. It will then return to the starting position. The procedure will be repeated for both legs.
Popliteal angle test | Baseline
  In the supine position, the hip and knee will be brought to 90 degrees. The digital inclinometer will be placed on the tuberositas tibia and the participant will be asked to extend the knee while maintaining the position of the hip. At the last point, the value on the inclinometer will be recorded. It will then return to the starting position. The procedure will be repeated for both legs.
Popliteal angle test | 1 hour
  In the supine position, the hip and knee will be brought to 90 degrees. The digital inclinometer will be placed on the tuberositas tibia and the participant will be asked to extend the knee while maintaining the position of the hip. At the last point, the value on the inclinometer will be recorded. It will then return to the starting position. The procedure will be repeated for both legs.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

REFERENCES:
- [Derived] Erol E, Bulut BN. Acute effect of instrument-assisted soft tissue mobilization on hamstring flexibility via fascial chain. BMC Musculoskelet Disord. 2024 Dec 19;25(1):1046. doi: 10.1186/s12891-024-08182-7. PMID 39702162